CLINICAL TRIAL: NCT01373255
Title: Balloon Catheter for Occlusion of the Pelvic Vasculature as an Adjuvant Therapy in Cases of Placenta Accreta
Brief Title: Balloon Catheters in Cases of Abnormal Placentation
Acronym: Accreta
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HaEmek Medical Center, Israel (Other)
Responsible Party: Principal Investigator, Raed Salim, MD, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0043-08-EMC; Acreta02 (Other: Emek Medical Center)
Record Dates: First submitted 2011-06-10; First posted 2011-06-14 (Estimated); Last update posted 2015-06-16 (Estimated); Status verified 2015-06

CONDITIONS: Post Partum Bleeding
Keywords: Placenta accreta; Internal iliac artery catheterization; Post partum bleeding
MeSH Terms: conditions — Postpartum Hemorrhage; Placenta Accreta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- internal iliac catheterization (Experimental): Women in this arm will undergo internal iliac artery catheterization prior to the cesarean delivery
  Interventions: Procedure: internal iliac catheterization
- No intervention (No Intervention): no intervention prior to cesarean

INTERVENTIONS:
Procedure: internal iliac catheterization — Women in this arm will undergo internal iliac artery catheterization prior to the cesarean delivery
  Other Names: internal iliac artery catheterization
  Arms: internal iliac catheterization

SUMMARY:
Placenta accreta is a relatively rare event, in which the placenta is abnormally implanted into the uterine myometrium. The most significant complication is intense bleeding, mainly during labor. The most important risk factors are previous cesarean delivery, placenta previa, and advanced maternal age. Cesarean hysterectomy is the recommended management. During the recent years, inserting intravascular balloon catheter for occlusion and/or arterial embolization, was introduced as an adjuvant therapy in order to minimize blood loss during cesarean hysterectomy or in conduct with conservative management with the intent of avoiding hysterectomy in selective cases. Contradicting reports exist regarding the effectiveness and safety of the catheters in cases of placenta accreta. The objective of this study is to estimate the efficacy of the balloon catheters among women diagnosed with a placenta accreta.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women age 18-45
* antepartum diagnosis of placenta accreta

Exclusion Criteria:

- women who refuse to participate

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Number of blood products transfused | 5 years

SECONDARY OUTCOMES:
Need for hysterectomy | 5 years
catheter's side effects | 5 years
Length of hospitalization | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Raed Salim, Principal Investigator — Dep. OB/GYN, HaEmek Medical Center, Afula, Israel
Locations (1):
- Haemek Medical Center, Afula, Israel

REFERENCES:
- [Derived] Salim R, Chulski A, Romano S, Garmi G, Rudin M, Shalev E. Precesarean Prophylactic Balloon Catheters for Suspected Placenta Accreta: A Randomized Controlled Trial. Obstet Gynecol. 2015 Nov;126(5):1022-1028. doi: 10.1097/AOG.0000000000001113. PMID 26444128